CLINICAL TRIAL: NCT03189095
Title: Project Workout on Wheels Internet Intervention (WOWii): Summative Evaluation With Randomized Clinical Trial
Brief Title: Workout on Wheels Internet Intervention (WOWii)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 016-093
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injuries
Keywords: exercise; physical activity; SCI; spinal cord injury; online
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: The investigators opted to use a wait-list control group to serve as an untreated comparison for the experimental group. From the investigators' perspective, people calling about an exercise trial want to receive an intervention, and thus, they believe it would be unethical to deny access to the intervention. Control group participants will be asked to continue their current activity level over the 16 weeks and following their posttest, they will be invited to participate in the WOWii program in full. The investigators will examine whether differential dropouts occur between those assigned to the experimental and wait-list control groups. The investigators previous exercise study conducted among women with mobility impairment indicated slightly lower attrition in the wait list control group, with no significant differences between those who withdrew and those who remained in the study by six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: WOWii (Workout on Wheels Internet Intervention)
- Wait-List Control (No Intervention)

INTERVENTIONS:
Behavioral: WOWii (Workout on Wheels Internet Intervention) — Participants will self-monitor their exercise on the WOWii website, which has a page to record the type, duration, and intensity of daily exercise bouts.
  Two devices will track participants' exercise, a Polar heart rate monitor (RS300X, Polar®), which will provide data on the day, duration, and intensity (average and maximum) of aerobic activity and an ActiGraph accelerometer (model GT3X), which detects movement in three planes to indicate frequency and intensity of movement throughout the day. Experimental participants will be provided a Polar heart rate monitor to wear during each exercise bout for the entire length of the 6-month study, and exercise data will be collected weekly.
  Physiological outcomes on fitness will be assessed by measuring weight and aerobic capacity in a Cardiopulmonary Lab by a doctoral-trained physical therapist.
  Participants will complete surveys to report on their exercise self-efficacy and perceived barriers.
  Arms: Intervention

SUMMARY:
Project WOWii examines how useful and effective an online format is for helping people with SCI get more exercise over 4 months. Study participants will meet over Skype weekly for 16 weeks and work through weekly online modules to start and stick with an accessible and individualized exercise program. Participants will be compensated for their time to attend fitness testing and complete surveys before and just after the 16-week program.

DETAILED DESCRIPTION:
This study will gather empirical evidence of the effectiveness of WOWii intervention in promoting changes in exercise behavior, fitness, and perceptions of exercise over the 16 week intervention as well as 2 months later for individuals living with SCI. The study staff will assess effectiveness by measuring participants (a) time spent each week doing aerobic exercise by self-report and objective monitoring, (b) aerobic capacity to assess fitness changes, and (c) self-reported perceptions of exercise barriers and self-efficacy at baseline, 4 months, and 6 months.

Participants will be randomly assigned to an experimental (WOWii) or a wait-list control group in one of four cohorts over a two-year period. This was an effective strategy in our previous trial in helping us achieve the full sample size. We will use a blocked randomization procedure to assure equal distribution of those with paraplegia and tetraplegia. Four cohorts will be enrolled over two years, with each having up to 36 people. This allows for up to 18 participants in the experimental and control groups, which permits us to offer two different time options for participants to attend the weekly meetings, as our video conferencing software allows up to 10 people to participate in the group video chat. Each cohort will be divided into two groups of 18 study participants as experimental and wait-list control groups. The experimental group will be divided into two groups of nine participants. Each cohort will begin the intervention at the same time and attend weekly calls together. All participants will undergo a pre-screen assessment which includes eligibility assessment. Participants will undergo 2 in-person fitness testing assessments at baseline at the end of the 16 week internet intervention with online meetings, before or during which they will complete an online survey and follow. A third follow up assessment will be conducted as an online survey at 6 months, which is 2 months after the intervention is complete, and an exit survey will be conducted individually over the phone after within one week of completing the final online survey. The wait-list control group will be offered the intervention at the end of the 6 month period. Due to low enrollment numbers, we will likely add a 5th cohort for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 - 70 years old;
* Have SCI > 6 months with the ability to use arms enough for arm-based exercise and requires wheelchair use;
* Have access to a computer with internet access or if they do not have computer/internet access, have experience using a computer and going online;
* Obtain physician signed approval to participate in the exercise study; and
* Not be currently physically active, based on responses to the 7-item Behavioral Risk Factor Surveillance physical activity survey.

Exclusion Criteria:

* Not receive physician approval to begin an exercise program;
* Have participated in the previous pilot studies; and
* Unable to read the English language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in aerobic exercise (Participant adoption) | 16 weeks
  minutes per week measured by Polar activity tracker (objective)
Aerobic exercise maintenance | 16 weeks
  minutes per week measured by Polar activity tracker (objective)
Change in aerobic exercise (Participant adoption) | Baseline & 16 weeks
  minutes per week measured by The International Physical Activity Questionnaire (IPAQ) (subjective)
Aerobic exercise maintenance | 16 weeks
  minutes per week measured by The International Physical Activity Questionnaire (IPAQ) (subjective)

SECONDARY OUTCOMES:
Change in aerobic fitness | Baseline & 16 weeks
  peak V02 using continuous, graded arm crank protocol
Exercise Self-Efficacy | 16 weeks
  health promotion scale with exercise subscale Self Rated Abilities for Health Practices Scale (SRAHP)
Change in perceived exercise barriers | Baseline & 16 weeks
  Change in summary score of barriers on The Barriers to Health Activities among Disabled Persons scale (BHADP) from baseline to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Froehlich-Grobe, Ph.D., Principal Investigator — Baylor Institute for Rehabilitation
Locations (1):
- Baylor Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No